CLINICAL TRIAL: NCT04760119
Title: Drug-Eluting Balloon Angioplasty Versus Bypass Surgery as First-Line Strategies in Infrageniculate Arterial Disease for Critical Limb Ischemia in Type 2 Diabetic Pacients: a Randomised Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Viktoras Šliaužys, M.D., Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS3005
Record Dates: First submitted 2021-01-22; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: The treatment will consist of two treatment modalities: 1) Vein bypass surgery first strategy; 2) Endovascular treatment first (drug coated balloon angioplasty) strategy
Masking Description: Blinding is not possible due to the completely different natures of the treatments allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vein bypass surgery first strategy (Active Comparator)
  Interventions: Procedure: Vein bypass surgery first strategy
- Endovascular treatment first (drug coated balloon angioplasty) strategy (Active Comparator)
  Interventions: Procedure: Endovascular treatment first (drug coated balloon angioplasty) strategy

INTERVENTIONS:
Procedure: Vein bypass surgery first strategy — Vein bypass will be performed with standart anaesthetic and surgical techniques using reversed great saphenous vein conduit. Location of proximal and distal anastomosis will be recorded. Post surgery completion angiography imaging will be performed.
  Arms: Vein bypass surgery first strategy
Procedure: Endovascular treatment first (drug coated balloon angioplasty) strategy — Endovascular treatment using drug-coated balloons will be performed under local anaesthetic via common femoral artery. Final angiography imaging will be demonstrated.
  Arms: Endovascular treatment first (drug coated balloon angioplasty) strategy

SUMMARY:
The aim of this study is to evaluate the outcomes of drug-eluting balloon angioplasty and vein bypass surgery in diabetic patients with critical limb ischemia due to infrapopliteal arterial disease.

DETAILED DESCRIPTION:
Objective: To consider the clinical outcomes of drug-coated ballon angioplasty and vein bypass surgery in terms of amputation-free survival, overall survival, relief of symptoms, quality of life and to determine if limb revascularization contributes to diabetic peripheral neuropathy (DPN).

All patients with type 2 diabetes mellitus and severe limb ischemia reffered to multidisciplinary diabetic foot team or endocrinology or vascular units can be considered.

To be eligible for randomization, peripheral arterial occlusive disease must be located infra-popliteally; patients must have adequate inflow and outflow to support infrapopliteal interventions; have a good superficial vein for bypass surgery. If the patient is suitable for both treatment arms, they will be invited to enter the trial.

If patient is suitable for both revascularization techniques randomization will be performed after diagnostic angiogram submission

Patient will be randomised to one of the following groups:

A. Vein bypass surgery first strategy B. Endovascular treatment first (drug coated balloon angioplasty) strategy

Outcomes will be recorded at 1, 3, 6, 9, 12, 18, 24 month after revascularisation procedure. Information collected will include further interventions (vascular, non-vascular), hospitalisations (for whatever reason), other health problems, clinical and haemodinamic status of limbs, funcional status, quality of life, neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 2 diabetes mellitus
* Severe limb ischemia (Rutherford class >=4) due to infrapopliteal, +/- popliteal disease [ a.tibialis anterior, tr.tibioperonealis, a.peronea, a.tibialis posterior, a.dorsalis pedis stenosis or occlusion (50%-100%; >40mm in length); leasion may involve a.poplitea P1-P3 segment; have adequate inflow and outflow to support infrapopliteal intervention (diagnostic imaging); suitable for both vein bypass and best endovascular treatment following; angiography diagnostic imaging and ultrasound examination of vein conduit.]

Exclusion Criteria:

* Requires primary limb amputation
* Acute limb ischemia
* Anticipated life expectancy of <2 years
* Unsuitable for either revascularisation strategy
* Severe concomitant disease (acute coronary ischemic event, brain ischemic event, cognitive disorder, active oncology process)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary, primary-assisted and secondary patency | 24 months
  Clinical and ultrasound assesment

SECONDARY OUTCOMES:
Ischemic symptoms | 24 months
  Fontaine classification: I asymptomatic; IIa mild claudication; IIb moderate-to-severe claudication; III rest pain; IV ulceration or gangrene.
  Rutherford classification: 0 asymptomatic; 1 mild claudication; 2 moderate claudication; 3 severe claudication; 4 rest pain; 5 minor tissue loss; 6 severe tissue loss or gangrene.
Ankle-brachial index (ABI) | 24 months
  Ratio of the blood pressure at the ankle to the blood pressure in the upper arm. Norm 1.0-1.4
Toe-brachial index (TBI) | 24 months
  Ratio of the blood pressure of the great toe to the blood pressure in the upper arm. Norm 1.0-1.4
Transcutaneous oxygen tension (TcPO2) | 24 months
  A noninvasive test that directly measures the oxygen level of tissue beneath the skin. A TcPO2 greater than 55 mmHg is considered normal regardless of the site of measurement, whereas a value of 40 mmHg is the critical value below which wound healing is impaired and ischemia develops.
Healing of tissue loss (ulcers, gangrene) | 24 months
  Clinical examination and photo documentation.
Re- and cross-over intervention rates | 24 months
Major and minor amputation rates | 24 months
In-hospital morbidity/mortality and overall survival | 24 months
Relief of pain: Visual analog scale (VAS) | 24 months
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain).
Quality of life: EQ-5D-5L questionaire | 24 months
  Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension.
Diabetic neuropathy dinamics: clinical examination of foot sensation | 24 months
  Full hypoesthesia; Partial hypoesthesia; No changes; + Assymetry.
Diabetic neuropathy dinamics: neurometer | 24 months
  Perception threshold measurement. Neurometer® determines three sub-types of nerve fiber by producing transcutaneous electrical stimuli at frequencies of 2000, 250 and 5 Hz.
Diabetic neuropathy dinamics: electroneuromiography | 24 months
  Diagnostic procedure that evaluates the health condition of muscles and the nerve cells that control them. A nerve conduction velocity between 50 and 60 meters per second is generally considered in the normal range.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, LT, Lithuania

IPD SHARING:
Plan to Share IPD: No